CLINICAL TRIAL: NCT01447940
Title: Prospective Assessment of Meos Telemedicine E-portal on Ambulatory Care of Type 1 Diabetic Patients
Acronym: TELEDIAB-3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DCIC10 20
Record Dates: First submitted 2011-10-03; First posted 2011-10-06 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Telemedicine; Type 1 diabetes; economic cost of Type 1 diabetes; ePortal Meos
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Care (Placebo Comparator): Patients will have conventional care with 2 standard visits (inclusion and 12 months) + HbA1c measure at 6 months. Patients won't use Meos ePortal
  Interventions: Device: Meos ePortal use
- Meos ePortal use (Experimental): Patients will use Meos ePortal + 2 standard visits (inclusion and 12 months) + additional visits if necessary + HbA1c measure at 6 months
  Interventions: Device: Meos ePortal use

INTERVENTIONS:
Device: Meos ePortal use — Patients will use Meos ePortal + 2 standard visits (inclusion and 12 months) + additional visits if necessary + HbA1c measure at 6 months
  Other Names: Telemedicine; ePortal

SUMMARY:
Primary objective of TELEDIAB-3 study is to demonstrate that the use of Meos Telemedicine ePortal for sharing information between diabetologist and type 1 diabetic patient is not inferior to a conventional care regarding metabolic results at 12 months.

DETAILED DESCRIPTION:
Meos is the name of the website (Telemedicine ePortal) tested in this trial ; it is used to share informations between diabetologist and type 1 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 1 diabetes mellitus for ≥ 12 months or more
* Age > 18 years old
* Patient who is followed since 6 month into investigator hospital
* Patient with available internet access at least once a week, and ability to understand MEOS website navigation
* Patient using a compatible glucose meter (One touch ultra, Optium xceed, or BG star)

Exclusion Criteria:

* Patient with no easy and regular access to the Internet;
* Patient found to be unfit for use of the telematic tools or e-mail tools
* Patient with toxicomania, alcoholism or psychological troubles
* Type 2 diabetic patients
* Patient who does not need strict metabolic objectives
* Pregnant or parturient women
* Person with no freedom (prisoner)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c measured at 12 months in Meos ePoral group versus conventional care group. Non-inferiority level is defined at a 0.15% threshold for an expected HbA1c of 8.5% at 12 months | 12 months

SECONDARY OUTCOMES:
HbA1c measured at 6 months in each group | 6 months
HbA1c measured at 12 months in each group | 12 months
HbA1c measured at 6 months in each group according to initial HbA1c level (higher than 8% or to median) | 6 months
HbA1c measured at 12 months in each group according to initial HbA1c level (higher than 8% or to median) | 12 months
Definition of failure: study withdraws or emergency hospitalization linked to diabetes or HbA1c increase of 0.5 % up to 12 months of follow up | 12 months
Annual cost of diabetes care from hospital and health insurance' points of view | 12 months
Quality of life at inclusion and 12 months, using the Diabetes Health Profile (DHP-1) scale and the Satisfaction items of the Diabetes Quality of Life (DQOL) questionnaire | 12 months
Qualitative analysis by semi-structured interviews, then quantitative survey by questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Benhamou, Pr, Principal Investigator — University Hospital, Grenoble
Locations (8):
- France (8):
  - University Hospital, Department of Endocrinology, Grenoble, Auvergne-Rhône-Alpes
  - University Hospital of Caen (Hospital Côte de nacre), Caen, Basse-Normandie
  - University Hospital of Besancon - Hospital Jean Minjoz, Besançon, Franche Comté
  - Hospital University of Montpellier, Montpellier, Languedoc-Roussillon
  - University Hospital of Reims, Reims, Marne
  - University Hospital of Nantes, Nantes, Pays de la Loire Region
  - University Hospital of Lyon (HCL Lyon sud), Lyon, Rhônes-Alpes
  - Hospital Sud Francilien, Corbeil Essonne, Île-de-France Region

REFERENCES:
- [Background] Chase HP, Pearson JA, Wightman C, Roberts MD, Oderberg AD, Garg SK. Modem transmission of glucose values reduces the costs and need for clinic visits. Diabetes Care. 2003 May;26(5):1475-9. doi: 10.2337/diacare.26.5.1475. PMID 12716807
- [Background] Farmer AJ, Gibson OJ, Dudley C, Bryden K, Hayton PM, Tarassenko L, Neil A. A randomized controlled trial of the effect of real-time telemedicine support on glycemic control in young adults with type 1 diabetes (ISRCTN 46889446). Diabetes Care. 2005 Nov;28(11):2697-702. doi: 10.2337/diacare.28.11.2697. PMID 16249542
- [Background] Montori VM, Helgemoe PK, Guyatt GH, Dean DS, Leung TW, Smith SA, Kudva YC. Telecare for patients with type 1 diabetes and inadequate glycemic control: a randomized controlled trial and meta-analysis. Diabetes Care. 2004 May;27(5):1088-94. doi: 10.2337/diacare.27.5.1088. PMID 15111526
- [Background] Benhamou PY, Melki V, Boizel R, Perreal F, Quesada JL, Bessieres-Lacombe S, Bosson JL, Halimi S, Hanaire H. One-year efficacy and safety of Web-based follow-up using cellular phone in type 1 diabetic patients under insulin pump therapy: the PumpNet study. Diabetes Metab. 2007 Jun;33(3):220-6. doi: 10.1016/j.diabet.2007.01.002. Epub 2007 Mar 28. PMID 17395516
- [Background] Boizel R, Benhamou PY, Renard E; Accu-Chek Pocket Compass Study Group. Glucose monitoring and pump data management software operated on a personal digital assistant can contribute to improve diabetes control in CSII-treated patients. Diabetes Metab. 2007 Sep;33(4):314-5. doi: 10.1016/j.diabet.2007.03.001. Epub 2007 May 1. No abstract available. PMID 17475533
- [Background] Young RJ, Taylor J, Friede T, Hollis S, Mason JM, Lee P, Burns E, Long AF, Gambling T, New JP, Gibson JM. Pro-active call center treatment support (PACCTS) to improve glucose control in type 2 diabetes: a randomized controlled trial. Diabetes Care. 2005 Feb;28(2):278-82. doi: 10.2337/diacare.28.2.278. PMID 15677779
- [Background] Ralston JD, Revere D, Robins LS, Goldberg HI. Patients' experience with a diabetes support programme based on an interactive electronic medical record: qualitative study. BMJ. 2004 May 15;328(7449):1159. doi: 10.1136/bmj.328.7449.1159. PMID 15142919
- [Background] Cho JH, Chang SA, Kwon HS, Choi YH, Ko SH, Moon SD, Yoo SJ, Song KH, Son HS, Kim HS, Lee WC, Cha BY, Son HY, Yoon KH. Long-term effect of the Internet-based glucose monitoring system on HbA1c reduction and glucose stability: a 30-month follow-up study for diabetes management with a ubiquitous medical care system. Diabetes Care. 2006 Dec;29(12):2625-31. doi: 10.2337/dc05-2371. PMID 17130195
- [Background] Tate DF, Jackvony EH, Wing RR. Effects of Internet behavioral counseling on weight loss in adults at risk for type 2 diabetes: a randomized trial. JAMA. 2003 Apr 9;289(14):1833-6. doi: 10.1001/jama.289.14.1833. PMID 12684363
- [Background] Trief PM, Sandberg J, Izquierdo R, Morin PC, Shea S, Brittain R, Feldhousen EB, Weinstock RS. Diabetes management assisted by telemedicine: patient perspectives. Telemed J E Health. 2008 Sep;14(7):647-55. doi: 10.1089/tmj.2007.0107. PMID 18817493